CLINICAL TRIAL: NCT04351399
Title: Psychological Impact of Quarantine in Rheumatoid Arthritis Patient During COVID-19 Outbreak
Acronym: PRPsyCOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_29; 2020-A00907-32 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-04

CONDITIONS: Sars-CoV2; Rheumatic Diseases; Rheumatoid Arthritis; Chronic Pain
Keywords: Psychological impact; COVID-19; Rheumatoid arthritis
MeSH Terms: conditions — Rheumatic Diseases; Arthritis, Rheumatoid; Chronic Pain; COVID-19

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with chronic painful inflammatory rheumatism
  Interventions: Other: questionnaire assesment

INTERVENTIONS:
Other: questionnaire assesment — The questionnaire will ask questions around their socio-demographic characteristics,quality of life, painful, using analgesic , since they are in quarantine

SUMMARY:
Clinical data about psychological impact of quarantine are well studied in transient event or more prolonged situation like jail incarceration.

In recent metaanalysis, psychological impact of quarantine was well documented in a specific population during first SARS epidemy. Even after the end of quarantine several patients were still with symptom of avoiding mainly agoraphobia, frequent hand washing and a carefull return to normal life COVID-19 infection is already associated with psychological symptom like anxiety, depression, sleep disorders and symptoms of acute stress However psychological impact of quarantine is on none in chronic painful inflammatory rheumatism in France. The prevalence of rheumatoid arthritis is 0.5% of the population with frequent comorbidity such as anxiety and depression.

During the quarantine secondary to COVID-19 pandemic it's possible to evaluated the psychological impact of adult RA patients.

The present study is an "emergency" being realize before the end of the quarantine.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis Quarantine

Exclusion Criteria:

* Non adult patient RA patient without quarantine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA patient will be interviewed par internet questionnaire (patient association / ANDAR)
Sampling Method: Non-Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Frequency of RA patients with emotional impact (feeling of isolation) | maximum 1 week from baseline on

SECONDARY OUTCOMES:
self-reported questionnaire for painful | maximum 1 week from baseline on
  Self reported questionnaire with questions to assess the characteristic,intensity of pain on quality of life, and consumption of analgesic.

CONTACTS AND LOCATIONS:
Overall Officials: René-Marc FLIPO, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hopital Roger Salengro, CHU Lille, Lille, France